CLINICAL TRIAL: NCT03908515
Title: Multi-center Clinical Observation of FCVB in Guangdong Province
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Xiaofeng Lin, associate dean of Zhongshan Ophthalmic Center, Sun Yat-sen University, Sun Yat-sen University
Other Study IDs: FCVB 2019
Record Dates: First submitted 2019-04-05; First posted 2019-04-09 (Actual); Last update posted 2019-04-16 (Actual); Status verified 2019-04

CONDITIONS: Retina Detachment; Eye Injuries; Eye Atrophy; Silicone Emulsion
Keywords: Foldable Capsular Vitreous Body; Retina detachment; eye atrophy
MeSH Terms: conditions — Retinal Detachment; Eye Injuries

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Foldable Capsular Vitreous Body (FCVB) — FCVB can be regarded as an artificial vitreous and consists of a thin vitreous-shaped capsule, a drain tube, and a valve. After foldable implantation into the eye, then silicone oil is injected into the capsule which inflated to support the retina. The capsular material of FCVB is silicone rubber. The capsule was fabricated a computer simulation of the human and rabbit vitreous cavities. The control of the intraocular pressure is achieved with adjusting the amount of injected medium through the tube-valve system. After the medium was injected into the capsule through the tube-valve system, the valve was subsequently fixed onto the sclera surface similar to the glaucoma valve.

SUMMARY:
This study provides further theoretical guidance for clinical application of FCVB through observing and collecting various indicators before and after surgical treatment of the FCVB in the real world.

DETAILED DESCRIPTION:
1. Research purpose: Collect and analyze the medical data in clinical work, in order to provide further theoretical guidance for the clinical application of FCVB.
2. Inclusion criteria: 1) Patients with severe retinal detachment, cannot be cured with existing vitreous substitutes, and are scheduled for FCVB implantation surgery; 2) Patients with silicone oil dependent eye, silicone oil emulsification, and chooses FCVB surgery; 3) Patients whose eyeball Atrophy, and strongly demand eye protection.
3. Exclusion criteria: 1) Patients with positive urine pregnancy test; 2) Patients with FCVB removed and switched to other alternative treatments; 3) Patients the investigator consider are not suitable for this clinical trial.
4. Endpoint Primary endpoint: Changes in corneal transverse diameter and ocular protrusion after 1 year of FCVB implantation.

   Secondary endpoints: visual acuity and intraocular pressure; local inflammatory response and complications evaluation; satisfaction investigated by questionnaire survey.
5. Process Before surgery, collecting the patient's medical history and pre-operative related specialist examination data and subjective opinions of doctors on surgical indications. Recording the surgical procedure, intraoperative complications. After surgery (3 days, 1 week, 2 weeks, 4 weeks, 3 months, 6 months after surgery, 1 year and 1 year follow-up every year), using visual acuity chart, slit lamp microscope, ophthalmoscope, intraocular pressure, Hertel exophthalmometer, vernier caliper to observe the patient's visual acuity, local inflammatory reaction, intraocular pressure and eyeball atrophy changes.
6. Efficacy evaluation Main indicators: the changes of corneal transverse diameter and ocular protrusion were observed 1 year after FCVB implantation.

   Secondary indicators: visual acuity and intraocular pressure; local inflammatory response and complications evaluation; satisfaction investigated through questionnaire survey.
7. Safety evaluation Adverse events that occurred during all studies.
8. Termination criteria During the clinical trial, the clinical trial shall be terminated in any of the following cases; (1) FCVB cannot be implanted (2) Subjects who fail to comply with the program requirements (including loss of follow-up) are subject to termination by the study physician; (3) a female patient who is intentionally pregnant or a female subject who has been confirmed to have been pregnant; (4) Participated in other clinical trials after participating in this clinical trial; (5) Adverse events or serious adverse events occurred during the trial and were unable to continue participating in the study; (6) The subject withdraws the informed consent or requests termination of the trial for some objective reason.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with the diagnose that severe retinal detachment and cannot be cured with existing vitreous substitutes, or silicone oil dependent eye accompanied with silicone oil emulsification, or eyeball atrophy meanwhile patients strongly demand keeping eyeball.
2. Patients agree to receive FCVB implantation surgery.

Exclusion Criteria:

1. Patients whose urine pregnancy test are positive.
2. Patients whose FCVB have been removed and switched to other alternative treatments.
3. Patients whom the investigator consider are not suitable for this clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients are scheduled for FCVB implantation surgery
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2019-05-01 (Estimated); Primary Completion 2019-05-31 (Estimated); Study Completion 2020-05-31 (Estimated)

PRIMARY OUTCOMES:
Corneal transverse diameter change | Corneal transverse diameter change from 1day before surgery to 1 year after surgery
  Determine the degree of eyeball atrophy through the change of transverse Diameter of the cornea
Ocular protrusion change | Ocular protrusion change from 1day before surgery to 1 year after surgery
  Determine the degree of eyeball atrophy through the ocular protrusion change

SECONDARY OUTCOMES:
Visual acuity | 3 days, 1 week, 2 weeks, 4 weeks, 3 months, 6 months after surgery, 1 year after surgery
  Postoperative visual acuity
Intraocular pressure | 3 days, 1 week, 2 weeks, 4 weeks, 3 months, 6 months after surgery, 1 year after surgery
  Postoperative intraocular pressure
Local inflammatory response | 3 days, 1 week, 2 weeks, 4 weeks, 3 months, 6 months after surgery, 1 year after surgery
  Evaluation of postoperative complications
Patients satisfaction | 3 days, 1 week, 2 weeks, 4 weeks, 3 months, 6 months after surgery, 1 year after surgery
  Postoperative patients satisfaction

CONTACTS AND LOCATIONS:
Overall Officials: Xiaofeng Lin, PhD, Study Chair — Zhongshan Ophthalmic Center, Sun Yat-sen University
Locations (1):
- Zhongshan Ophthalmic Center of Sun yat-sen Universtiy, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No